CLINICAL TRIAL: NCT03119142
Title: Economic Crisis and Adherence to the Mediterranean Diet: Possible Impact on Biomarkers of Inflammation and Metabolic Phenotypes in the Cohort of the MOLI-SANI Study
Brief Title: Economic Crisis and Adherence to the Mediterranean Diet (CASSIOPEA)
Acronym: CASSIOPEA
Status: Completed | Type: Observational
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Marialaura Bonaccio, PhD, Neuromed IRCCS
Other Study IDs: 5/17
Record Dates: First submitted 2017-04-10; First posted 2017-04-18 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Dietary Habits; Inflammation; Economic Problems; Obesity; Diabetes; Hypertension
MeSH Terms: conditions — Feeding Behavior; Inflammation; Obesity; Diabetes Mellitus; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Blood samples will be obtained from participants who had fasted overnight and had refrained from smoking for at least 6 h and stored in liquid nitrogen in the Biological bank of the Moli-sani study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The socioeconomic gradient in health is well known and is partially explained by differences in health-related behaviours across socioeconomic groups. There is reason to believe that the current economic crisis has been contributing to the observed rapid decrease in the adherence to the Mediterranean diet, thus reducing a protective factor against the development of major chronic diseases. This project aims at investigating whether the economic crisis could account for the shifting from the Mediterranean diet. Additionally, it will address variations in inflammation biomarkers (possibly dietary-related) or metabolic phenotypes as useful biological accounts for the decline in the adherence to Mediterranean diet. This project will also test whether for economically weakest people cultural resources could somehow attenuate the impact of material circumstances on lifestyle changes attributable to the economic crisis.

DETAILED DESCRIPTION:
Specific aims:

Aim 1: To identify population groups differently affected by the economic crisis within the population-based cohort of the MOLI-SANI study recruited in the years 2005-2006 (before economic crisis). This aim will be achieved by a new assessment of self-reported economic difficulties possibly emerged after the recruitment.

Aim 2: To estimate possible changes in dietary and health-related behaviours (with particular focus on the adherence to the Mediterranean diet) in subjects identified in the previous aim as highly or poorly affected by the economic crisis. Inflammatory status and metabolic phenotypes will be assessed in the two groups, recalled in a suitable proportion, to establish a possible link between shifting from the Mediterranean diet and adverse health outcomes. Quality of life and stress status will also be evaluated.

Aim 3: To evaluate in the group more affected by economic constraints whether nutrition knowledge and mass media exposure would account for the decline in the adherence to the Mediterranean diet and consequent changes in inflammatory status and/ or metabolic phenotypes.

Experimental Design Aim 1: Aim 1 will identify two groups of subjects as being most or less affected by the economic crisis. This aim will be reached by recall of 7,000 individuals from the Moli-sani cohort recruited in the years 2005-2006. Subjects will be administered a questionnaire to assess economic constraints likely occurred after the economic crisis onset. The questionnaire will update socioeconomic position and estimate economic constraints, food quality and food expenditure.

Experimental Design Aim 2: Within the two groups identified in aim 1, aim 2 will:

1. Perform a dietary follow up by administering the Italian version of the EPIC questionnaire (9), already used at baseline, to estimate the changes in dietary habits. Lifestyle follow up will be obtained by a validated questionnaire used at baseline.
2. Assess changes in inflammatory status by measurements of the following biomarkers: High-sensitivity C-reactive protein, Interleukin-6, Interleukin-18, Tumor necrosis factor, Plasminogen activator inhibitor-1, VCAM, ICAM, P-selectin, E-selectin, L-selectin, CD40L, adiponectin, platelet and leukocyte counts, lipids, triglycerides, glucose, insulin.
3. Estimate variations in the metabolic phenotypes (prevalence of hypertension, diabetes, obesity, metabolic syndrome, and levels of blood pressure, hip and waist circumferences).

Experimental Design Aim 3: A validated questionnaire on nutrition knowledge and exposure to mass media will be administered. This will allow to retrospectively identify additional subgroups differently exposed to information in order to estimate the role of cultural resources in health-related behavioural changes.

ELIGIBILITY:
Inclusion Criteria:

* The present study will include subjects recruited in the Moli-sani cohort during 2005-2006 and for which inclusion criteria were:
* aged >=35 years
* inscribed in the city hall registries

Exclusion Criteria:

* The present study will include subjects recruited in the Moli-sani cohort during 2005-2006 and for which exclusion criteria were:
* pregnancy at the time of recruitment,
* disturbances in understanding or willingness
* current poly-traumas or coma, refusal to sign the Informed Consent form

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MOLI-SANI is a population-based cohort study that recruited, between 2005 and 2010, 24,325 men and women at random from individuals aged 35 years or older resident in the Molise region, to investigate genetic and environmental risk factors for cardiovascular, cerebrovascular and tumour diseases. Of them, the present study will include about 7,000 subjects recruited in 2005-2006.
Sampling Method: Probability Sample
Enrollment: 3646 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Adherence to the Mediterranean diet | The follow-up is of 10 years since baseline enrolment (2005-2010)
  Dietary information will be collected by administering the Italian version of the EPIC questionnaire (Pala V et al. Tumori. 2003;89:594-607), already used at baseline, to estimate the changes in dietary habits. Adherence to a Mediterranean dietary pattern will be evaluated both by a priori (Mediterranean Diet Score; Trichopoulou A et al. N Engl J Med. 2003;348:2599-608) and a posteriori approach (Principal Factor Analysis; Centritto F et al. Nutr Metab Cardiovasc Dis. 2009;19:697-706).

SECONDARY OUTCOMES:
Obesity | The follow-up is of 10 years since baseline enrolment (2005-2010)
  Body mass index (BMI) will be obtained by dividing weight in kilograms (kg) by height (meters) squared. Obesity will be defined according to the following BMI categories: Underweight = <18.5; Normal weight = 18.5-24.9; Overweight = 25-29.9; Obesity = BMI of 30 or greater.
Hypertension | The follow-up is of 10 years since baseline enrolment (2005-2010)
  Hypertension will be defined as systolic blood pressure ≥140 mm Hg or diastolic blood pressure ≥90 mm Hg or treatment for hypertension.
Hypercholesterolemia | The follow-up is of 10 years since baseline enrolment (2005-2010)
  Hypercholesterolemia will be defined if total cholesterol ≥240 mg/dl or by use of specific medication.
Diabetes | The follow-up is of 10 years since baseline enrolment (2005-2010)
  Diabetes will be defined as blood glucose ≥126 mg/dl or by use of specific pharmacological treatment.
Inflammation | The follow-up is of 10 years since baseline enrolment (2005-2010)
  Inflammatory status will be assessed by measurements of the following biomarkers: High-sensitivity C-reactive protein, Interleukin-6, Interleukin-18, Tumor necrosis factor, Plasminogen activator inhibitor-1, VCAM, ICAM, P-selectin, E-selectin, L-selectin, CD40L, adiponectin, platelet and leukocyte counts, lipids, triglycerides, glucose, insulin.

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs Neuromed, Campobasso, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bonaccio M, Costanzo S, Di Castelnuovo A, Persichillo M, De Curtis A, Olivieri M, Cerletti C, Donati MB, de Gaetano G, Iacoviello L; CASSIOPEA Study and Moli-sani Study Investigators. The CASSIOPEA Study (Economic Crisis and Adherence to the Mediterranean diet: poSSIble impact on biOmarkers of inflammation and metabolic PhEnotypes in the cohort of the Moli-sAni Study): Rationale, design and characteristics of participants. Nutr Metab Cardiovasc Dis. 2021 Apr 9;31(4):1053-1062. doi: 10.1016/j.numecd.2020.12.008. Epub 2020 Dec 13. PMID 33549444